CLINICAL TRIAL: NCT06722716
Title: Study of Pneumococcal Carriage in RSV Bronchiolitis in Infants Aged 6 to 18 Months
Acronym: Synergy
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Pneumococcal Reference Center (Unknown); Infectious Diseases Models for Innovative Therapies (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP240862; 2024-A01592-45 (Other: ANSM : Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-09-25; First posted 2024-12-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-08

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; pneumonia
MeSH Terms: conditions — Bronchiolitis; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bronchiolitis group: Nasopharyngeal swab
  Interventions: Other: Swab collection
- healthy group: Infants without RSV bronchiolitis
  Interventions: Other: Swab collection

INTERVENTIONS:
Other: Swab collection — Nasopharyngeal swab

SUMMARY:
The relationship between RSV (human respiratory syncytial virus) infections and invasive infections or pneumonia caused by Streptococcus pneumoniae has been observed epidemiologically for several years. Few fundamental data exist to support the epidemiological relationship. This study will investigate the proportion of pneumococcal carriage in RSV-infected infants and noninfected infants (proportion, serotype profile).

DETAILED DESCRIPTION:
The relationship between RSV (human respiratory syncytial virus) infections and Streptococcus pneumoniae pneumonia has been suggested for many years based on a similar seasonal pattern and cohort studies, but it could not be confirmed due to the circulation of several viruses concurrently. The post-COVID-19 period was marked by a temporal association between RSV infections and invasive pneumococcal disease (and pneumonia) in children under five, highlighting the potential role of RSV in the dynamics of pneumococcal disease in infants.

Furthermore, the carriage rate of S. pneumoniae in infants under 2 years of age in healthy populations is described as around 25%. In the case of RSV infection, this rate rises to 50%. Some data from animal models have shown that RSV infection increases S. pneumoniae transmission within a group of individuals, partly explaining this difference. However, data remain limited, particularly in human samples, and further research is needed to better understand the role of the RSV-pneumococcal relationship in the occurrence of severe RSV infections (pneumonia) and invasive pneumococcal infections. This study will examine pneumococcal carriage in bronchiolitis in infants aged 6-18 months, through nasopharyngeal swabs from infants with bronchiolitis and healthy infants. Pneumococcal carriage rates and serotype profiles will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 6 months to 18 months inclusive
* With bronchiolitis during RSV epidemic season (bronchiolitis group) or without evidence of RSV viral infection (healthy group)
* No chronic illness
* No history of bronchiolitis
* Signed consent from parents or legal guardians
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Chronic respiratory illness
* Medical history of bronchiolitis or newborn asthma
* Treatment with immunosuppressants
* Patient on AME

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The included population will consist of infants aged 6 to 18 months, divided into two groups. On one hand, infants with RSV bronchiolitis (regardless of severity) and on the other hand, RSV-negative infants (consulting for other reasons, such as trauma, jaundice, etc.). The recruitment age is justified by the peak occurrence of invasive pneumococcal infections, which typically occurs around 12 months of age.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
nasopharyngeal carriage rate of Streptococcus pneumoniae (Sp) | Inclusion
  Comparison of nasopharyngeal carriage rates of Streptococcus pneumoniae (Sp) in healthy infants and infants with RSV bronchiolitis.

SECONDARY OUTCOMES:
serotype profile | Inclusion
  Comparison of the predominant serotype between the two groups.
serotype profile | Inclusion
  Comparison of the distribution of each serotype between the two groups.
proportion of 13-valent and 23-valent vaccine serotypes | Inclusion
  the proportion of 13-valent and 23-valent vaccine serotypes among pneumococcal strains between the two groups
proportion of non-vaccine serotypes | Inclusion
  proportion of non-vaccine serotypes among all pneumococcal strains between the two groups
Serotype profile distribution | Inclusion
  Serotypic Profile (Distribution of Serotypes) of S. pneumoniae in Nirsevimab-treated versus non-treated infants under 12 months of age, as assessed by nasopharyngeal swabs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Antoine Béclère, Clamart, France